CLINICAL TRIAL: NCT00003344
Title: Phase I-II Study of Weekly CPT-11 and Radiation Therapy for Unresectable or Locally Recurrent Large Bowel Cancer
Brief Title: Radiation Therapy Plus Irinotecan in Treating Patients With Colon Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Purpose: Treatment
Other Study IDs: CDR0000066321; MUSC-7532; HCC/MUSC-GI-01; NCI-V98-1420
Record Dates: First submitted 1999-11-01; First posted 2004-09-13 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Colorectal Cancer
Keywords: stage II colon cancer; stage III colon cancer; stage II rectal cancer; stage III rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Irinotecan; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: irinotecan hydrochloride
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining radiation therapy with chemotherapy may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of radiation therapy plus irinotecan in treating patients with colon cancer that is recurrent or that cannot be removed surgically.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose (MTD) of weekly irinotecan that will result in an acceptable level of toxicity when given in combination with concurrent external beam radiation therapy. II. Determine the objective response rate of these patients at the dose level below the MTD.

OUTLINE: Patients receive irinotecan IV over 90 minutes beginning within 24 hours of radiotherapy on days 1, 8, 15, and 22. External beam radiotherapy is administered 5 days per week for 5.5-6 weeks starting on day 1 concurrent with chemotherapy. Cohorts of 3-6 patients are treated until the maximum tolerated dose (MTD) has been determined. The MTD is defined as the dose level at which the incidence of dose limiting toxicity is no greater than one-third of the patients treated at that dose level. Once the MTD has been determined, additional patients receive irinotecan at the dose level below the MTD with external beam radiation therapy on the same treatment schedule as above. Patients are followed at 4 weeks after treatment, then every 3 months for 2 years, and then every 6 months for 3 additional years.

PROJECTED ACCRUAL: Approximately 3-24 patients will be accrued into the Phase I portion of this study. Approximately 15-25 patients will be accrued into the Phase II portion of this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed unresectable, incompletely resected with gross residual disease, or locally recurrent large bowel carcinoma confined to a site within the abdomen or pelvis All disease must be encompassable within a single radiotherapy port No evidence of uncontrolled metastatic disease outside of the planned radiotherapy port

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: CALGB 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 2.0 mg/dL Renal: Not specified Cardiovascular: No history of significant myocardial disease No New York Heart Association class III or IV disease No unstable angina No myocardial infarction in the past 4 months Other: No significant infection or other coexistent medical condition that would preclude protocol therapy Maintain an adequate oral nutrition intake (at least 1,200 calories estimated per day) No greater than 6 bowel movements per day prior to treatment No significant nausea or emesis on optimal antiemetic therapy Not pregnant or nursing Effective contraception required of all fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior irinotecan Endocrine therapy: Not specified Radiotherapy: No prior abdominal or pelvic radiotherapy Surgery: At least 3 weeks since laparotomy or laparoscopic procedure with or without resection

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49
Dates: Start 1998-08; Primary Completion 2000-01 (Actual); Study Completion 2000-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles R. Thomas, MD, Study Chair — The University of Texas Health Science Center at San Antonio
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States